CLINICAL TRIAL: NCT04707534
Title: Effects of Higher Dose and Lower Dose of Dexamethasone for Hospitalized Patients With COVID-19
Brief Title: Comparing the Effects of Different Doses of Dexamethasone to Treat Inpatient COVID-19
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12927
Record Dates: First submitted 2021-01-11; First posted 2021-01-13 (Actual); Results first posted 2024-03-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Covid19
Keywords: COVID 19
MeSH Terms: conditions — COVID-19 | interventions — Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexamethasone 20 mg (Experimental): Dexamethasone 20 mg daily for 5 days, followed by dexamethasone 10 mg daily for 5 days
  Interventions: Drug: Dexamethasone
- Dexamethasone 6 mg (Active Comparator): Dexamethasone 6 mg daily for 10 days
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone

SUMMARY:
This open label clinical trial is to evaluate two different doses of dexamethasone on the health outcome using World Health Organization ordinal scale at day 28 in hospitalized patients with COVID-19.

DETAILED DESCRIPTION:
The coronavirus disease 2019 (COVID-19) pandemic is a serious global health threat. Multiple antiviral or immunomodulatory therapies have failed to show any mortality benefit for patients with COVID-19. Dexamethasone was shown in prior studies to improve mortality and ventilator free days. However, it is unclear what dose of dexamethasone is most beneficial in hospitalized patients with COVID-19. This randomized single center open label clinical trial is to evaluate two different doses of dexamethasone (20mg vs. 6mg) on the health outcome for hospitalized patients with COVID-19. The intervention arm is dexamethasone 20mg daily for 5 days, followed by dexamethasone 10mg daily for 5 days. The comparator is dexamethasone 6mg daily for 10 days. Three hundred participants will be enrolled. The primary outcome is clinical improvement using World Health Organization ordinal scale at day 28.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* RT-PCR confirmed COVID-19 infection
* Positive pressure ventilation (non-invasive or invasive) or high flow nasal cannula (HFNC) or need supplemental oxygen with oxygen mask or nasal cannula

Exclusion Criteria:

* Underlying disease requiring chronic corticosteroids
* Severe adverse events before admission, i.e. cardiac arrest;
* Contraindication for corticosteroids;
* Death is deemed to be imminent and inevitable during the next 24 hours
* Recruited in other clinical intervention trial
* Pregnancy
* Patient on judicial protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2021-01-21 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Huimin Wu, MD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Medical Center, Oklahoma City, Oklahoma, United States

REFERENCES:
- [Derived] Wu H, Daouk S, Kebbe J, Chaudry F, Harper J, Brown B. Low-dose versus high-dose dexamethasone for hospitalized patients with COVID-19 pneumonia: A randomized clinical trial. PLoS One. 2022 Oct 3;17(10):e0275217. doi: 10.1371/journal.pone.0275217. eCollection 2022. PMID 36190994

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dexamethasone 20 mg | Dexamethasone 6 mg
Started | 55 | 55
Dexamethasone 20mg | 52 | 0
Dexamethasone 6mg | 0 | 55
Completed | 52 | 55
Not Completed | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexamethasone 20 mg | Dexamethasone 6 mg | Total
Number analyzed (Participants) | 52 | 55 | 107
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (14) | 58 (17) | 57 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 26 | 51
  Male | 27 | 29 | 56
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 4
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 17 | 32
  White | 29 | 24 | 53
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 5 | 10 | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Improvement of Greater Than or Equal to 2 Points Using the WHO-OSCI at Day 28
Description: the clinical improvement of greater than or equal to 2 points using the WHO-OSCI. 1. Not hospitalized, no limitations on activities 2. Not hospitalized, limitation on activities 3. Hospitalized, not requiring supplemental oxygen 4. Hospitalized, requiring supplemental oxygen by mask or nasal prongs 5. Hospitalized, on non-invasive ventilation or high flow oxygen devices 6. Hospitalized, on invasive mechanical ventilation 7. Hospitalized, on invasive mechanical ventilation + additional organ support (pressors, RRT, ECMO) 8. Death
Time Frame: 28 days from study enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone 20 mg | Dexamethasone 6 mg
Number analyzed (Participants) | 52 | 55
Participants | 37 | 43

2. Secondary Outcome: 28-day Mortality
Description: All-cause mortality at 28 days after enrollment
Time Frame: 28 days from study enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone 20 mg | Dexamethasone 6 mg
Number analyzed (Participants) | 52 | 55
Participants | 11 | 5

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | Dexamethasone 20 mg | Dexamethasone 6 mg
All-Cause Mortality (participants affected / at risk) | 11/52 | 5/55
Serious Adverse Events (participants affected / at risk) | 1/52 | 2/55
Other Adverse Events (participants affected / at risk) | 6/52 | 10/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dexamethasone 20 mg (N=52) | Dexamethasone 6 mg (N=55)
Ventilator associated pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dexamethasone 20 mg (N=52) | Dexamethasone 6 mg (N=55)
hyperglycemia, requires insulin infusion (Endocrine disorders) | 2 | 1
bacteremia (Infections and infestations) | 3 | 10
Catheter-related bloodstream infection (Infections and infestations) | 1 | 3
Candidemia (Infections and infestations) | 0 | 1
Pulmonary aspergillosis (Infections and infestations) | 0 | 1
Gastrointestinal bleeding (Gastrointestinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-15): https://cdn.clinicaltrials.gov/large-docs/34/NCT04707534/Prot_SAP_000.pdf